CLINICAL TRIAL: NCT00827632
Title: Oral Contraception and Ovarian Suppression in Women With Different Weights
Brief Title: Obesity, Oral Contraception, and Ovarian Suppression
Acronym: 20/30
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carolyn L. Westhoff, Professor of Obstetrics and Gynecology, Population and Family Health and Epidemiology at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAB4823; R01HD045786 (NIH)
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Suppression
Keywords: Ovarian Suppression; Oral Contraceptives; Obese and Normal BMI
MeSH Terms: conditions — Obesity | interventions — Dosage Forms; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Weight group (Active Comparator): Participants with a BMI of 19-24.9 kg/m^2
  Interventions: Drug: Low dose formulation; Drug: High dose formulation
- Obese group (Active Comparator): Participants with a BMI of 30-39.9 kg/m^2
  Interventions: Drug: Low dose formulation; Drug: High dose formulation

INTERVENTIONS:
Drug: Low dose formulation — Participants are randomized to either Portia (levonorgestrel/ethinyl estradiol tablets, United States Pharmacopeia (USP)0.15 mg/0.03 mg or Lessina (levonorgestrel/ethinyl estradiol tablets, USP 0.1 mg/0.02 mg) for 3 months use.
  Dose formula contains 20 ug of ethinyl estradiol (EE) and 100 ug of levonorgestrel (LN) per tablet.
  Other Names: Low dose
Drug: High dose formulation — Participants are randomized to either Portia (levonorgestrel/ethinyl estradiol tablets, United States Pharmacopeia (USP)0.15 mg/0.03 mg or Lessina (levonorgestrel/ethinyl estradiol tablets, USP 0.1 mg/0.02 mg) for 3 months use.
  Dose formula contains 30 ug of ethinyl estradiol (EE) and 150 ug of levonorgestrel (LN) per tablet.
  Other Names: High dose

SUMMARY:
This study proposes a double blind randomized clinical trial to include normal weight and obese women who have normal ovulatory function at baseline; the investigators will randomize women to 2 widely used OCs and evaluate ovarian follicle development and circulating progesterone to assess ovarian suppression during OC use.

DETAILED DESCRIPTION:
There is a large gap between lowest expected failure rates of about 1.5% and typical use failure rates of about 7% per year. This gap may be due to incorrect use or to decreased oral contraceptive (OC) effectiveness in population subgroups. Recent reports suggest greater OC failure among heavier women, particularly those using the lowest doses. The prevalence of obesity in the US population has recently increased to about 23% in women aged 20-29, peak years for OC use. OC physiology and effectiveness have not been evaluated in obese women.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35
* Body Mass Index (BMI) 19-24.9 or 30-39.9 kg/m^2
* Willing to take birth control pills for 3-4 months
* Recent spontaneous pregnancy or cyclic menses

Exclusion Criteria:

* Contraindications to hormonal contraceptives
* Oophorectomy/Polycystic ovary syndrome (PCOS)
* Taken oral contraceptives to regulate menses recently
* Weight reduction surgery
* Used Depo-Provera within the last 12 months
* Pregnant or currently breastfeeding
* Desiring pregnancy within the next 4 months
* Unable to make study visit commitment
* Previous participation in this study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Mayeda ER, Torgal AH, Westhoff CL. Weight and body composition changes during oral contraceptive use in obese and normal weight women. J Womens Health (Larchmt). 2014 Jan;23(1):38-43. doi: 10.1089/jwh.2012.4241. Epub 2013 Oct 24. PMID 24156617
- [Derived] Westhoff CL, Torgal AH, Mayeda ER, Stanczyk FZ, Lerner JP, Benn EKT, Paik M. Ovarian suppression in normal-weight and obese women during oral contraceptive use: a randomized controlled trial. Obstet Gynecol. 2010 Aug;116(2 Pt 1):275-283. doi: 10.1097/AOG.0b013e3181e79440. PMID 20664386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant-related activities were conducted between July 2006-December 2008 in New York City
Pre-assignment Details: Eligible women were aged 18-35 years with a recent history of regular, spontaneous menstrual cycles, and agreed to use an Oral Contraceptive Pill (OCP) for 3 to 4 months and undergo eight biweekly study visits during the third or fourth OCP cycle.
Groups:
- Normal Weight: Participants with a Body Mass Index (BMI) of 19-24.9.
- Obese: Participants with a Body Mass Index (BMI) of 30-39.9.
Period: Overall Study
Arm/Group | Normal Weight | Obese
Started | 128 | 98
Completed | 106 | 75
Not Completed | 22 | 23
Not completed — Lost to Follow-up | 8 | 12
Not completed — Early withdrawal | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Weight | Obese | Total
Number analyzed (Participants) | 106 | 75 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 106 | 75 | 181
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 75 | 181
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 19 | 19 | 38
  Non-Hispanic African American | 30 | 23 | 53
  Non-Hispanic White | 33 | 11 | 44
  Non-Hispanic Asian | 14 | 1 | 15
  Non-compliant OCP users (dropped from analysis) | 10 | 21 | 31
Oral Contraceptive Pill Compliance [Number; unit: Participants]
  Consistent Users | 96 | 54 | 150
  Inconsistent Users | 4 | 9 | 13
  Nonusers | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Risk of Oral Contraceptive (OC) Failure Due to Less Contraceptive-mediated Ovarian Suppression.
Description: Perpendicular diameter, ethinyl estradiol, and progesterone values were used to create Hoogland Scores. Hoogland Scores were used to assess ovarian suppression during OC use. The Hoogland Score comprises 6 grades (Because of small numbers, grades 5 and 6 were combined):
  1. no activity
  2. potential activity
  3. nonactive follicle-like structure
  4. active follicle-like structure
  5. luteinized unruptured follicle
  6. ovulation
  Each participant received a score from 1-6 to indicate the level of ovarian suppression; total number of participants were tallied for each Hoogland score.
Time Frame: Up to 8 biweekly visits from start of OCP therapy
Population: Two hundred twenty-six women enrolled, 150 consistent OCP users were retained for the main analysis (96 normal weight and 54 obese).
Measure: Number; unit: Participants
Arm/Group | Normal Weight | Obese
Number analyzed (Participants) | 96 | 54
Participants
  Score of 1 - no activity | 54 | 28
  Score of 2 - potential activity | 11 | 12
  Score of 3 - nonactive follicle-like structure | 6 | 6
  Score of 4 - active follicle-like structure | 21 | 7
  Score of 5/6 - luteinization or ovulation | 4 | 1

2. Secondary Outcome: Lipid or Carbohydrate Metabolism in Obese Versus Normal Weight Oral Contraceptive (OC) Users at Baseline and Exit Visit (12-16 Weeks OC Exposure).
Time Frame: Screening (baseline) and follow-up 1 (exit)
Population: We excluded participants who were not compliant with the study treatment (based on measuring serum hormone concentrations) from the analyses.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Normal Weight | Obese
Number analyzed (Participants) | 96 | 54
mg/dL
  Baseline Carbohydrate - Glucose | 87.2 (8.6) | 90.2 (7.1)
  Exit Carbohydrate - Glucose | 89.8 (8.5) | 92.7 (10.5)
  Baseline Lipid - Total Cholesterol | 171.4 (25.9) | 177.0 (27.2)
  Exit Lipid - Total Cholesterol | 172.3 (27.3) | 170.4 (35.8)

3. Secondary Outcome: Pharmacokinetics of 15 Obese Weight and 15 Normal Weight Women on Combined Oral Contraceptives.
Time Frame: 24 hours during week 3 of follow-up cycle
Population: Data were not available. No analysis performed.
Arm/Group | Normal Weight | Obese
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Normal Weight | Obese
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/54
Other Adverse Events (participants affected / at risk) | 0/96 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No